CLINICAL TRIAL: NCT03998163
Title: An Open-Label, Multicenter Study to Evaluate the Safety and Effectiveness of Intravenous CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus
Brief Title: CR845-CLIN3105: A Study to Evaluate the Safety and Effectiveness of CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR845-CLIN3105
Record Dates: First submitted 2019-05-07; First posted 2019-06-26 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Uremic Pruritus
Keywords: Hemodialysis; Pruritus; Uremic Pruritus; Dialysis; CR845; Chronic Itch; CKD; CKD-associated pruritus; CKD-aP; ESRD (end stage renal disease); difelikefalin; Itch; Itching; KALM; Chronic Kidney Disease; Kidney failure, chronic; Kidney dysfunction; Generalized pruritus
MeSH Terms: conditions — Pruritus; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — difelikefalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CR845 0.5mcg/kg (Experimental): IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
  Interventions: Drug: CR845 0.5 mcg/kg

INTERVENTIONS:
Drug: CR845 0.5 mcg/kg — IV CR845 0.5 mcg/kg administered three times/week
  Other Names: CR845; Difelikefalin

SUMMARY:
This is a multicenter, open-label study to evaluate the safety and effectiveness of intravenous (IV) CR845 at a dose of 0.5 mcg/kg administered after each dialysis session. The study includes an up to 12-week Treatment Period.

DETAILED DESCRIPTION:
Screening Period: The Screening Period includes a Screening Visit and a Run-In Period. Informed consent will be obtained prior to performing any study-specific procedures. The Screening Visit will occur within 21 days prior to the start of the Run-in Period. Patients will start the Run-in Period during the week prior to Treatment Period to complete eligibility verification.

Treatment Period: All scheduled study visits during the Treatment Period will be conducted on dialysis days. Patients will be administered CR845 as an IV bolus after the end of their dialysis during a Treatment Period of up to 12 weeks so that each patient will receive CR845 3 times weekly for a total of up to 36 doses. End of treatment (EOT) is defined as the first day of dialysis following the last dose of drug. The EOT procedures will be conducted on the dialysis visit following the last dose of study drug.

Follow-up Visit: A final safety Follow up Visit will be conducted 7-10 days after the EOT/Early Termination Visit.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* Has end-stage renal disease (ESRD) and has been on hemodialysis 3 times per week for at least 3 months prior to the start of screening;
* Has at least 2 single-pool Kt/V measurements ≥1.2, or at least 2 urea reduction ratio measurements ≥65%, or 1 single pool Kt/V measurement ≥1.2 and 1 urea reduction ratio measurement ≥65% on different dialysis days during the 3 months period prior to screening;
* Prior to Treatment:

  * Has completed at least 3 Worst Itching Intensity NRS questionnaires from the start of the Run-in Period up to and including the pre-dose assessment on Day 1;

Key Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Known noncompliance with dialysis treatment that in the opinion of the investigator would impede completion or validity of the study;
* Scheduled to receive a kidney transplant during the study;
* New or change of treatment received for itch including antihistamines and corticosteroids (oral, IV, or topical) within 14 days prior to screening;
* New or change of prescription for opioids, gabapentin, or pregabalin within 14 days prior to screening;
* Received another investigational drug within 30 days or five half-lives (whichever is longer) prior to the start of dosing or is planning to participate in another interventional clinical study while enrolled in this study;
* Has pruritus only during the dialysis session (by patient report);
* Is receiving ongoing ultraviolet B treatment and/or anticipates receiving such treatment during the study;
* Participated in a previous clinical study with CR845.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (47):
- United States (33):
  - Cara Therapeutics Study Site, Escondido, California
  - Cara Therapeutics Study Site, Riverside, California
  - Cara Therapeutics Study Site, San Diego, California
  - Cara Therapeutics Study Site, Victorville, California
  - Cara Therapeutics Study Site, Denver, Colorado
  - Cara Therapeutics Study Site, Middlebury, Connecticut
  - Cara Therapeutics Study Site, Norwich, Connecticut
  - Cara Therapeutics Study Site, Coral Gables, Florida
  - Cara Therapeutics Study Site, Fort Lauderdale, Florida
  - Cara Therapeutics Study Site, Hollywood, Florida
  - Cara Therapeutics Study Site, Miami, Florida
  - Cara Therapeutics Study Site 2, Tampa, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Albany, Georgia
  - Cara Therapeutics Study Site, Boston, Massachusetts
  - Cara Therapeutics Study Site, Roseville, Michigan
  - Cara Therapeutics Study Site, Minneapolis, Minnesota
  - Cara Therapeutics Study Site, Kansas City, Missouri
  - Cara Therapeutics Study Site, Las Vegas, Nevada
  - Cara Therapeutics Study Site 2, Las Vegas, Nevada
  - Cara Therapeutics Study Site, Great Neck, New York
  - Cara Therapeutics Study Site, Philadelphia, Pennsylvania
  - Cara Therapeutics Study Site, Spartanburg, South Carolina
  - Cara Therapeutics Study Site, Knoxville, Tennessee
  - Cara Therapeutics Study Site, Austin, Texas
  - Cara Therapeutics Study Site, Duncanville, Texas
  - Cara Therapeutics Study Site, Greenville, Texas
  - Cara Therapeutics Study Site, Mansfield, Texas
  - Cara Therapeutics Study Site, Mesquite, Texas
  - Cara Therapeutics Study Site 2, San Antonio, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site 3, San Antonio, Texas
  - Cara Therapeutics Study Site, Temple, Texas
- Czechia (4):
  - Cara Therapeutics Study Site, Havlíčkův Brod
  - Cara Therapeutics Study Site, Nové Město na Moravě
  - Cara Therapeutics Study Site, Prague
  - Cara Therapeutics Study Site, Sokolov
- Hungary (7):
  - Cara Therapeutics Study Site 2, Budapest
  - Cara Therapeutics Study Site, Budapest
  - Cara Therapeutics Study Site, Dunaújváros
  - Cara Therapeutics Study Site, Kaposvár
  - Cara Therapeutics Study Site, Kistarcsa
  - Cara Therapeutics Study Site, Nyíregyháza
  - Cara Therapeutics Study Site, Szombathely
- Poland (3):
  - Cara Therapeutics Study Site, Ostrołęka
  - Cara Therapeutics Study Site, Radom
  - Cara Therapeutics Study Site, Sochaczew

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fishbane SN, Block GA, Evenepoel P, Budden J, Morin I, Menzaghi F, Wen W, Lerma EV. Pruritus Severity and Serum Phosphate in CKD: A Post Hoc Analysis of Difelikefalin Studies. Kidney360. 2024 Sep 1;5(9):1270-1280. doi: 10.34067/KID.0000000000000520. Epub 2024 Jul 22. PMID 39037824
- [Derived] Fotheringham J, Guest J, Latus J, Lerma E, Morin I, Schaufler T, Soro M, Stander S, Zeig S. Impact of Difelikefalin on the Health-Related Quality of Life of Haemodialysis Patients with Moderate-To-Severe Chronic Kidney Disease-Associated Pruritus: A Single-Arm Intervention Trial. Patient. 2024 Mar;17(2):203-213. doi: 10.1007/s40271-023-00668-1. Epub 2024 Jan 9. PMID 38196014
- [Derived] Weiner DE, Schaufler T, McCafferty K, Kalantar-Zadeh K, Germain M, Ruessmann D, Morin I, Menzaghi F, Wen W, Stander S. Difelikefalin improves itch-related sleep disruption in patients undergoing haemodialysis. Nephrol Dial Transplant. 2024 Jun 28;39(7):1125-1137. doi: 10.1093/ndt/gfad245. PMID 37968132
- [Derived] Weiner DE, Vervloet MG, Walpen S, Schaufler T, Munera C, Menzaghi F, Wen W, Bhaduri S, Germain MJ; trial investigators. Safety and Effectiveness of Difelikefalin in Patients With Moderate-to-Severe Pruritus Undergoing Hemodialysis: An Open-Label, Multicenter Study. Kidney Med. 2022 Aug 24;4(10):100542. doi: 10.1016/j.xkme.2022.100542. eCollection 2022 Oct. PMID 36185706
- [Derived] Fishbane S, Wen W, Munera C, Lin R, Bagal S, McCafferty K, Menzaghi F, Goncalves J. Safety and Tolerability of Difelikefalin for the Treatment of Moderate to Severe Pruritus in Hemodialysis Patients: Pooled Analysis From the Phase 3 Clinical Trial Program. Kidney Med. 2022 Jun 28;4(8):100513. doi: 10.1016/j.xkme.2022.100513. eCollection 2022 Aug. PMID 36039153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CR845 0.5mcg/kg
Started | 222
Completed | 197
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | CR845 0.5mcg/kg
Number analyzed (Participants) | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 110
  White | 96
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AEs.
Description: Assessed by monitoring of adverse events.
Time Frame: Up to Follow-Up Visit (Week 13-14)
Measure: Count of Participants; unit: Participants
Arm/Group | CR845 0.5mcg/kg
Number analyzed (Participants) | 222
Participants | 143

ADVERSE EVENTS:
Time Frame: Up to Follow-Up Visit (Week 13-14)
Arm/Group | CR845 0.5mcg/kg
All-Cause Mortality (participants affected / at risk) | 3/222
Serious Adverse Events (participants affected / at risk) | 45/222
Other Adverse Events (participants affected / at risk) | 11/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.5mcg/kg (N=222)
Anaemia (Blood and lymphatic system disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Chronic left ventricular failure (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Primary adrenal insufficiency (Endocrine disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Enterocoloitis (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Osteomyelitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1
Corynebacterium test positive (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5
Fluid overload (Metabolism and nutrition disorders) | 2
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hypertensive urgency (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.5mcg/kg (N=222)
Diarrhoea (Gastrointestinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT03998163/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT03998163/SAP_001.pdf